CLINICAL TRIAL: NCT01468090
Title: Risk of Surgery Among Patients Wih Ulcerative Colitis and Croh'ns Disease After Seven Years of Follow-up in the Era of Biological Treatment.
Brief Title: Disease Course in an IBD Cohort in the Era of Biological Treatment
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Ferring Pharmaceuticals (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Marianne Vester-Andersen, Principal investigator, Hvidovre University Hospital
Other Study IDs: 562_2003_2004
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Inflammatory bowel disease; Crohn's disease; Ulcerative colitis; Disease course; Phenotype; Biological treatment
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and faeces will be retained for biobank
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Disease course: 562 patients diagnosed with Crohn's disease (209), ulcerative colitis (326) or indeterminant colitis (27) in the period of 1st of January 2003 to 31st of December 2004 in Copenhagen City and County (an area covering 23% of the Danish population).

SUMMARY:
The aim of the study is to do a 7-year follow-up of a consecutive inception cohort of 562 adults and children diagnosed and registered with inflammatory bowel disease in 2003-04 in order to evaluate the consequences of biological therapy in the treatment of IBD. The cohort is established after the implementation of biological agents in the treatment of IBD and the investigators hypothesis is that a) Severe disease course in IBD can be predicted by phenotypic presentation by serological, genetic, clinical and endoscopic characteristics to be used as guidance in the selection of treatment strategy and b) Introduction of biological treatment changes the course of disease in IBD and reduces the need of surgical procedures.

Methods: Medical records will be reviewed to register the use of medication, flare ups (medical and surgical) and hospital admissions. Diagnosis, disease localization and behavior will be evaluated. At outpatient visits patients will get a clinical examination, blood and faeces will be collected to biobank and patients will be offered an endoscopical examination. The Montreal classification, The Harvey & Bradshaw's activity index (CD) and the SCAAI score (UC) will be used to describe disease localization, extent, behavior and severity. An electronic database will be established in use of processing data.

ELIGIBILITY:
Inclusion Criteria:

* All patients wil be followed up and diagnosis will be reassessed.

Exclusion Criteria:

* Non-IBD (after reassessing diagnosis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 562 patients diagnosed with Crohn's disease, Ulcerative colitis or indeterminant colitis in 2003-2004 i Copenhagen City and County and registered in a database.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Surgical rate | 7 years from inception (2003-04)
  The risk of intestinal surgery from inception (2003-04) until 7 years of follow-up in Crohn's disease and ulcerative colitis

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Vester-Andersen, MD, Principal Investigator — Dep. of Gastroenterology 360, Hvidovre Hospital; Pia Munkholm, MD, DMsc, Study Chair — Dep. of Gastroenterology, Herlev Hospital; Ida Vind, MD, PhD, Study Chair — Dep. of gastroenterology, Amager Hospital; Flemming Bendtsen, prof. DMsci, Study Director — Gastroenheden 360 Hvidovre University Hospital
Locations (2):
- Denmark (2):
  - Hvidovre Hospital, Gastroenheden 360, Hvidovre
  - Hvidovre hospital, Hvidovre